CLINICAL TRIAL: NCT04799886
Title: Attitudes Associated to Prescription of ADHD Drugs Among Child and Adolescent Psychiatrists in Region Skåne.
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: RSLUAFADHD2021
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Attitude; ADHD - Combined Type; Physician's Role
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Child and adolescent psychiatrist
  Interventions: Other: Semi structured interview

INTERVENTIONS:
Other: Semi structured interview — Interviews are performed by one research group member and based on beforehand decided questions and sub-questions. The interview material is transcribed and analysed on a theme level.

SUMMARY:
Each year Region Skåne in Sweden gathers information on drug prescriptions within the region. The last ten years a significant pattern of uneven prescription rates of ADHD drugs to people up to 17 years of age are noticed in the different districts. These regional differences are noticed in other regions in Sweden as well and internationally.

The convention on the rights of the child became an institutional law in Sweden in 2020 and it emphasises that each child has the right to equal care and treatment. Therefore it is of importance to analyse how the variations in prescriptions rates arise and if we as healthcare providers can influence it. Our study is a collaboration between Region Skåne and the university of Lund and is a part of a larger study of the regional variations of prescriptions of ADHD drugs. Previous research informs us that a complex interplay of multiple factors can be behind variations in prescription rates among medical doctors and not the least subjective experiences and attitudes.

Our study performs semistructured interviews of Region Skånes child and adolescent psychiatrists with questions specifically regarding their own experiences and attitudes that might influence their prescription behavior.

The intention is to gather information that can guide future research questions.

ELIGIBILITY:
Inclusion Criteria:

* child and adolescent psychiatrist in Region Skåne

Exclusion Criteria:

* part of the research group

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All child and adolescent psychiatrists in Region Skåne are informed about the study and ask for participation.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Attitudes and experiences associated with prescription and diagnosis of ADHD | 1 day (During the analysis of the transcribed interview)
  Semistructured interview

CONTACTS AND LOCATIONS:
Locations (1):
- Child and Adolescent Psychiatry, Region Skane, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mykletun A, Widding-Havneraas T, Chaulagain A, Lyhmann I, Bjelland I, Halmoy A, Elwert F, Butterworth P, Markussen S, Zachrisson HD, Rypdal K. Causal modelling of variation in clinical practice and long-term outcomes of ADHD using Norwegian registry data: the ADHD controversy project. BMJ Open. 2021 Jan 19;11(1):e041698. doi: 10.1136/bmjopen-2020-041698. PMID 33468528
- [Background] Zetts RM, Stoesz A, Garcia AM, Doctor JN, Gerber JS, Linder JA, Hyun DY. Primary care physicians' attitudes and perceptions towards antibiotic resistance and outpatient antibiotic stewardship in the USA: a qualitative study. BMJ Open. 2020 Jul 14;10(7):e034983. doi: 10.1136/bmjopen-2019-034983. PMID 32665343
- [Background] Fulton BD, Scheffler RM, Hinshaw SP, Levine P, Stone S, Brown TT, Modrek S. National variation of ADHD diagnostic prevalence and medication use: health care providers and education policies. Psychiatr Serv. 2009 Aug;60(8):1075-83. doi: 10.1176/ps.2009.60.8.1075. PMID 19648195
- [Background] Lindgren BM, Lundman B, Graneheim UH. Abstraction and interpretation during the qualitative content analysis process. Int J Nurs Stud. 2020 Aug;108:103632. doi: 10.1016/j.ijnurstu.2020.103632. Epub 2020 May 15. PMID 32505813